CLINICAL TRIAL: NCT04223570
Title: Portable Measurement of Protoporphyrin IX in the Skin
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Michael S. Chapman, Principal Investigator, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19167
Record Dates: First submitted 2019-12-24; First posted 2020-01-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-05

CONDITIONS: Photodynamic Therapy; Protoporphyrin IX
Keywords: Photodynamic Therapy; Actinic Keratoses; Protoporphyrin IX; Amino-levulinic acid
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Portable Apple Smart Phone Protoporphyrin IX Spectrometer Camera — This is a portable device that uses a camera to non-invasively and efficiently measure the level of protoporphyrin IX in various areas skin. This camera will be used in all participants to measure the level of protoporphyrin IX in various areas of skin as detailed in the study description.

SUMMARY:
Photodynamic therapy (PDT) is increasingly used to treat superficial skin lesions, such as actinic keratosis (AK) and non-melanoma skin cancers, and has been demonstrated to be an effective and safe alternative to surgery. It is performed by applying a photosensitizing pro-drug, amino -levulinic acid (ALA) and then allowing the conversion to the metabolite Protoporphyrin IX (PpIX). While attempts to measure the concentration of this drug in the skin have been performed before, there remains limited research on an individuals' baseline level of PpIX which could lead to the customization of PDT. With the development of a new handheld, smart phone-associated device to measure red fluoresce intensity of PpIX, this measurement is now feasible. This is an observational single center quantitative study in which the investigators will take measurements of red fluoresce intensity of PpIX at various locations. This will then be correlated with the individuals age, oral temperature, diet, and skin type. The investigators hypothesize that the levels of PpIX will depend on all of these factors, including anatomical location. All data will be collected into the data collection form and then analyzed. The investigators will assess for how anatomical location, skin pigmentation, oral temperature, and other factors influence PpIX levels. Fitzpatrick skin type will be assessed by the provider to assess skin pigmentation. All of these factors will be correlated to the PpIX levels in 5 anatomical locations (forehead, cheeks, forearms, hands, and bald scalp where applicable) to determine which factors most greatly influence the red fluoresce intensity of PpIX.

DETAILED DESCRIPTION:
Photodynamic Therapy (PDT) has gained popularity as an effective, non-scarring treatment for thin, non-hyperkeratotic actinic keratoses (AKs). Similar to the topical agents 5-fluorouracil and imiquimod, PDT is particularly useful when utilized as a field-directed therapy for the treatment of areas with multiple AKs and extensive sun damage. PDT consists of two steps: 1) the topical application of a photosensitizer agent aminolevulinic acid (ALA), which is preferentially converted to the photosensitive protoporphyrin IX (PpIX) in precancerous and neoplastic cells, and 2) controlled exposure to a visible wavelength light source. Current methodologies utilize a "one-size-fits-all" approach with regard to duration of incubation with photosensitizing agents and illumination. Moreover, patients frequently experience pain after long PDT prodrug incubation. Better characterization of photosensitization in PDT can help tailor incubation and overall treatment time to minimize treatment duration and discomfort while maximizing clearance of the target lesions. The direct measurement of PpIX is a promising, yet rarely performed test that may help determine the appropriate PDT treatment time, the need for re-treatment or adjuvant therapy, and potential efficacy of treatment. Point-probe measurements have shown extreme heterogeneity between PpIX levels in different patients and among different lesions in the same patient. However, these point-probe measurements are unable to account for the variance in PpIX production in different parts of the skin because of their relatively limited field of view. The recent development of a low-cost, smart phone-based, wide-field fluorescence dosimetry imaging system to map PpIX levels onto a 2D image allows for handheld, real-time analysis of PpIX levels in human skin. Initial unpublished clinical results have shown its utility in human subjects. However, a more extensive characterization of the factors that influence baseline in PpIX has yet to be performed. This study intends to elaborate these inter-and intra-individual variances, including analysis of changes in PpIX concentrations based on anatomical location, age, diet, temperature, pigmentation, and previous skin damage.

ELIGIBILITY:
Inclusion Criteria:

* All patients and staff appearing at the Dartmouth-Hitchcock Medical Center Heater Road Dermatology Clinic who are aged 18 years and older

Exclusion Criteria:

* Pregnant women
* Women who are breast-feeding
* Adults unable to consent
* Individuals who are not yet adults
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient subjects will be recruited at the DHMC outpatient dermatology clinic. Patients presenting for their routine sessions or regularly scheduled follow-up dermatology appointments will be provided information about the study. Employees at this location will also have the opportunity to participate.
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Protoporphyrin IX levels on the skin | At baseline
  Measure change in protoporphyrin IX levels in the skin of the forehead, malar cheek, dorsal hand, and dorsal forearm patients, as well as the bald scalp in male patients

SECONDARY OUTCOMES:
Effect of oral temperature on change in protoporphyrin IX levels at baseline and at serial time points after Ameluz application (the intervention) | At baseline
  Measure oral in temperature and compare it to protoporphyrin levels.
Effect of age on change in protoporphyrin IX levels at baseline and at serial time points after Ameluz application (the intervention) | At baseline
  Determine the relationship of participant age with change in protoporphyrin IX levels
Effect of Fitzpatrick skin type (skin pigmentation) on change in protoporphyrin IX levels | At baseline
  Determine the relationship of participant fitzpatrick skin type (skin pigmentation) with change in protoporphyrin IX levels
Effect of diet on change in protoporphyrin IX levels | At baseline
  Determine the relationship of participant diet with change in protoporphyrin IX levels
Effect of history of skin cancer on change in protoporphyrin IX levels | At baseline
  Determine the relationship of participant history of skin cancer with change in protoporphyrin IX levels
Effect of sex on change in protoporphyrin IX levels | At baseline
  Determine the relationship of participant sex with change in protoporphyrin IX levels

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Chapman, MD, MBA, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center Heater Road Clinic, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after being de-identified
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access these data.

REFERENCES:
- [Background] Landes R, Illanes A, Goeppner D, Gollnick H, Friebe M. A study of concentration changes of Protoporphyrin IX and Coproporphyrin III in mixed samples mimicking conditions inside cancer cells for Photodynamic Therapy. PLoS One. 2018 Aug 31;13(8):e0202349. doi: 10.1371/journal.pone.0202349. eCollection 2018. PMID 30169536
- [Background] Anand S, Ortel BJ, Pereira SP, Hasan T, Maytin EV. Biomodulatory approaches to photodynamic therapy for solid tumors. Cancer Lett. 2012 Dec 29;326(1):8-16. doi: 10.1016/j.canlet.2012.07.026. Epub 2012 Jul 25. PMID 22842096
- [Background] Tyrrell JS, Morton C, Campbell SM, Curnow A. Comparison of protoporphyrin IX accumulation and destruction during methylaminolevulinate photodynamic therapy of skin tumours located at acral and nonacral sites. Br J Dermatol. 2011 Jun;164(6):1362-8. doi: 10.1111/j.1365-2133.2011.10265.x. Epub 2011 May 13. PMID 21564050
- [Background] Kanick SC, Davis SC, Zhao Y, Hasan T, Maytin EV, Pogue BW, Chapman MS. Dual-channel red/blue fluorescence dosimetry with broadband reflectance spectroscopic correction measures protoporphyrin IX production during photodynamic therapy of actinic keratosis. J Biomed Opt. 2014;19(7):75002. doi: 10.1117/1.JBO.19.7.075002. PMID 24996661
- [Background] Nissen CV, Heerfordt IM, Wiegell SR, Mikkelsen CS, Wulf HC. Increased protoporphyrin IX accumulation does not improve the effect of photodynamic therapy for actinic keratosis: a randomized controlled trial. Br J Dermatol. 2017 May;176(5):1241-1246. doi: 10.1111/bjd.15098. Epub 2017 Mar 8. PMID 27696393
- [Background] Kanick SC, Davis SC, Zhao Y, Sheehan KL, Hasan T, Maytin EV, Pogue BW, Chapman MS. Pre-treatment protoporphyrin IX concentration in actinic keratosis lesions may be a predictive biomarker of response to aminolevulinic-acid based photodynamic therapy. Photodiagnosis Photodyn Ther. 2015 Dec;12(4):561-6. doi: 10.1016/j.pdpdt.2015.10.006. Epub 2015 Oct 22. PMID 26480810
- [Background] Nissen CV, Philipsen PA, Wulf HC. Protoporphyrin IX formation after topical application of methyl aminolaevulinate and BF-200 aminolaevulinic acid declines with age. Br J Dermatol. 2015 Sep;173(3):760-6. doi: 10.1111/bjd.13923. Epub 2015 Aug 20. PMID 25997508
- [Background] Zhao B, He YY. Recent advances in the prevention and treatment of skin cancer using photodynamic therapy. Expert Rev Anticancer Ther. 2010 Nov;10(11):1797-809. doi: 10.1586/era.10.154. PMID 21080805
- [Background] Alberto J. Ruiz, Ethan P. M. LaRochelle, M. Shane Chapman, Tayyaba Hasan, Brian Pogue. Smartphone-based fluorescence imager for PpIX-based PDT treatment planning: System design and initial results. In: Vol 10860. ; 2019. https://doi.org/10.1117/12.2510403.
- [Background] Rollakanti KR, Kanick SC, Davis SC, Pogue BW, Maytin EV. Techniques for fluorescence detection of protoporphyrin IX in skin cancers associated with photodynamic therapy. Photonics Lasers Med. 2013 Nov 1;2(4):287-303. doi: 10.1515/plm-2013-0030. PMID 25599015